CLINICAL TRIAL: NCT00807040
Title: Evaluation of Outcomes Following Mitral Valve Repair/Replacement in Severe Chronic Ischemic Mitral Regurgitation
Brief Title: Comparing the Effectiveness of Repairing Versus Replacing the Heart's Mitral Valve in People With Severe Chronic Ischemic Mitral Regurgitation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Alan Moskowitz, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 08-1078-00002; U01HL088942 (NIH); U01 HL088942-01-2; 595 (Other: Ct Surgery Network Research Group); NCT00919256 (obsolete NCT alias)
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Mitral Valve Insufficiency; Coronary Artery Disease
Keywords: Ischemic Mitral Regurgitation; Mitral Valve Disease; Severe Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mitral Valve Repair with Annuloplasty (Active Comparator): Participants will undergo mitral valve repair with annuloplasty and a sub-valvular procedure for severe tethering.
  Interventions: Procedure: Mitral Valve Repair with Annuloplasty
- Mitral Valve Replacement (Active Comparator): Participants will undergo mitral valve replacement and complete preservation of the sub-valvular apparatus.
  Interventions: Procedure: Mitral Valve Replacement

INTERVENTIONS:
Procedure: Mitral Valve Repair with Annuloplasty — The annuloplasty ring will be chosen by the surgeon. The ring is sized to the anterior leaflet and intertrigonal distance. A semi-rigid or rigid annuloplasty ring will be used, and if tethering is present, a subvalvar procedure will be performed.
  Arms: Mitral Valve Repair with Annuloplasty
Procedure: Mitral Valve Replacement — Mitral valve replacement will include complete preservation of the subvalvar apparatus. The technique of preservation, choice of prosthetic valve, and technique of suture placement will be dependent on the surgeon's preference. The prosthetic valve will be tested for paravalvular leaks by using the left ventricular saline infusion test.
  Arms: Mitral Valve Replacement

SUMMARY:
People with coronary artery disease (CAD) or people who have had a heart attack may develop a leak in the mitral valve of their heart and may therefore need to undergo surgery to fix the valve. The best way to fix the mitral valve remains undetermined. This study will evaluate whether it is better for people with severe mitral valve leakage to undergo a mitral valve replacement procedure or a mitral valve repair procedure.

DETAILED DESCRIPTION:
CAD occurs when the arteries that supply blood to the heart become blocked as a result of plaque buildup. In severe cases, CAD can cause chest pain, shortness of breath, and heart attack. After a heart attack, some people may develop a leak in the mitral valve of the heart. This condition is known as ischemic mitral regurgitation (IMR), and it can cause blood to flow backward into the heart. If left untreated, severe IMR can lead to heart failure or serious heart rhythm irregularities, known as arrhythmias. People with severe mitral valve leakage routinely undergo one of two surgical procedures to fix the mitral valve: a mitral valve repair procedure, in which a surgical ring is used to repair the valve; or a mitral valve replacement procedure, in which the damaged valve is replaced with a new one. Currently, there is no consensus in the medical community as to which procedure is more beneficial. The purpose of this study is to determine whether people with severe mitral valve regurgitation should undergo a mitral valve repair procedure or a mitral valve replacement procedure.

This study will enroll people with CAD who have severe mitral regurgitation. At a baseline study visit, participants will undergo a physical examination; blood collection; neurocognitive tests; and questionnaires regarding medical history, medication history, and quality of life. In the operating room, participants will be randomly assigned to undergo either the mitral valve repair procedure or the mitral valve replacement procedure. Blood, urine, and tissue samples may be collected from participants after the surgery; this is optional and will only be done with prior approval from participants. All participants will attend study visits at Day 30 and Months 6, 12, and 24. At each visit, participants will take part in a medication history review, a physical examination, an echocardiogram, a cardiopulmonary exercise test, neurocognitive tests, and quality of life surveys.

ELIGIBILITY:
Inclusion Criteria:

* Chronic severe ischemic mitral regurgitation (often with tethering as a major mechanism) in the judgment of the clinical site echocardiographer, assessed by transthoracic echocardiogram. Assessment of mitral regurgitation will be performed using an integrative method (Zoghbi W. et al. J. American Society of Echocardiography. 2003:16:777-802. see appendix). Quantitative guidelines as proposed would be: ERO ≥ 0.4 cmsq. If ERO < 0.4, then the degree of mitral regurgitation will be guided by other color Doppler quantitative methods (jet area/left atrial area ratio, vena contracta, supportive criteria in an integrated fashion
* Eligible for surgical repair and replacement of mitral valve
* CAD with or without the need for coronary revascularization

Exclusion Criteria:

* Any evidence of structural (chordal or leaflet) mitral valve disease or ruptured papillary muscle
* Prior mitral valve repair
* Severe irreversible pulmonary hypertension in the judgment of the investigator
* Medically unable to undergo cardiopulmonary bypass (CPB)
* Inability to derive ERO and end-systolic volume index (ESVI) by transthoracic echocardiography
* Planned concomitant intra-operative procedures (with the exception of tricuspid valve repair, closure of patent foramen ovale [PFO] or atrial septal defect [ASD] or Maze procedure)
* Clinical signs of cardiogenic shock at the time of surgery
* Treatment with long-term intravenous inotropic therapy at the time of surgery
* ST segment elevation myocardial infarction (MI) requiring intervention in the 7 days before surgery
* Congenital heart disease (except PFO or ASD)
* Evidence of cirrhosis or liver synthetic failure
* Excessive surgical risk, as judged by the surgical investigator
* Recent history of psychiatric disease (including drug or alcohol abuse) that is likely to impair compliance with the study, as judged by the investigator
* Therapy with an investigational intervention at the time of screening, or planning to enroll in an additional investigational intervention study during participation in this study
* Any concurrent disease with a life expectancy of less than 2 years
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2008-12; Primary Completion 2013-04 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Gardner, MD, Study Chair — Christiana Care Health Services; Patrick O'Gara, MD, Study Chair — Brigham and Women's Hospital; Annetine C. Gelijns, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (21):
- United States (18):
  - University of Southern California, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - University of Maryland, Baltimore, Maryland
  - NIH Heart Center at Suburban Hospital, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Montefiore Einstein Heart Center, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Duke University, Durham, North Carolina
  - East Carolina Heart Institute, Greenville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor Research Institute, Plano, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inova Heart and Vascular Institute, Falls Church, Virginia
- Canada (3):
  - Montreal Heart Institute, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - Quebec Heart Institute/Laval Hopital, Québec

REFERENCES:
- [Result] Acker MA, Parides MK, Perrault LP, Moskowitz AJ, Gelijns AC, Voisine P, Smith PK, Hung JW, Blackstone EH, Puskas JD, Argenziano M, Gammie JS, Mack M, Ascheim DD, Bagiella E, Moquete EG, Ferguson TB, Horvath KA, Geller NL, Miller MA, Woo YJ, D'Alessandro DA, Ailawadi G, Dagenais F, Gardner TJ, O'Gara PT, Michler RE, Kron IL; CTSN. Mitral-valve repair versus replacement for severe ischemic mitral regurgitation. N Engl J Med. 2014 Jan 2;370(1):23-32. doi: 10.1056/NEJMoa1312808. Epub 2013 Nov 18. PMID 24245543
- [Derived] Bertrand PB, Overbey JR, Zeng X, Levine RA, Ailawadi G, Acker MA, Smith PK, Thourani VH, Bagiella E, Miller MA, Gupta L, Mack MJ, Gillinov AM, Giustino G, Moskowitz AJ, Gelijns AC, Bowdish ME, O'Gara PT, Gammie JS, Hung J; Cardiothoracic Surgical Trials Network (CTSN). Progression of Tricuspid Regurgitation After Surgery for Ischemic Mitral Regurgitation. J Am Coll Cardiol. 2021 Feb 16;77(6):713-724. doi: 10.1016/j.jacc.2020.11.066. PMID 33573741
- [Derived] Giustino G, Overbey J, Taylor D, Ailawadi G, Kirkwood K, DeRose J, Gillinov MA, Dagenais F, Mayer ML, Moskowitz A, Bagiella E, Miller M, Grayburn P, Smith PK, Gelijns A, O'Gara P, Acker M, Lala A, Hung J. Sex-Based Differences in Outcomes After Mitral Valve Surgery for Severe Ischemic Mitral Regurgitation: From the Cardiothoracic Surgical Trials Network. JACC Heart Fail. 2019 Jun;7(6):481-490. doi: 10.1016/j.jchf.2019.03.001. PMID 31146872
- [Derived] Ferket BS, Ailawadi G, Gelijns AC, Acker M, Hohmann SF, Chang HL, Bouchard, D, Meltzer DO, Michler RE, Moquete EG, Voisine P, Mullen JC, Lala A, Mack MJ, Gillinov AM, Thourani VH, Miller MA, Gammie JS, Parides MK, Bagiella E, Smith RL, Smith PK, Hung JW, Gupta LN, Rose EA, O'Gara PT, Moskowitz AJ, Cardiothoracic Surgical Trials Network (CTSN) Investigators. Cost-Effectiveness of Mitral Valve Repair Versus Replacement for Severe Ischemic Mitral Regurgitation: A Randomized Clinical Trial From the Cardiothoracic Surgical Trials Network. Circ Cardiovasc Qual Outcomes. 2018 Nov 14;11(11):e004466. doi: 10.1161/CIRCOUTCOMES.117.004466. PMID 30785252
- [Derived] Capoulade R, Zeng X, Overbey JR, Ailawadi G, Alexander JH, Ascheim D, Bowdish M, Gelijns AC, Grayburn P, Kron IL, Levine RA, Mack MJ, Melnitchouk S, Michler RE, Mullen JC, O'Gara P, Parides MK, Smith P, Voisine P, Hung J; Cardiothoracic Surgical Trials Network (CTSN) Investigators. Impact of Left Ventricular to Mitral Valve Ring Mismatch on Recurrent Ischemic Mitral Regurgitation After Ring Annuloplasty. Circulation. 2016 Oct 25;134(17):1247-1256. doi: 10.1161/CIRCULATIONAHA.115.021014. PMID 27777294
- [Derived] Goldstein D, Moskowitz AJ, Gelijns AC, Ailawadi G, Parides MK, Perrault LP, Hung JW, Voisine P, Dagenais F, Gillinov AM, Thourani V, Argenziano M, Gammie JS, Mack M, Demers P, Atluri P, Rose EA, O'Sullivan K, Williams DL, Bagiella E, Michler RE, Weisel RD, Miller MA, Geller NL, Taddei-Peters WC, Smith PK, Moquete E, Overbey JR, Kron IL, O'Gara PT, Acker MA; CTSN. Two-Year Outcomes of Surgical Treatment of Severe Ischemic Mitral Regurgitation. N Engl J Med. 2016 Jan 28;374(4):344-53. doi: 10.1056/NEJMoa1512913. Epub 2015 Nov 9. PMID 26550689
- [Derived] Kron IL, Hung J, Overbey JR, Bouchard D, Gelijns AC, Moskowitz AJ, Voisine P, O'Gara PT, Argenziano M, Michler RE, Gillinov M, Puskas JD, Gammie JS, Mack MJ, Smith PK, Sai-Sudhakar C, Gardner TJ, Ailawadi G, Zeng X, O'Sullivan K, Parides MK, Swayze R, Thourani V, Rose EA, Perrault LP, Acker MA; CTSN Investigators. Predicting recurrent mitral regurgitation after mitral valve repair for severe ischemic mitral regurgitation. J Thorac Cardiovasc Surg. 2015 Mar;149(3):752-61.e1. doi: 10.1016/j.jtcvs.2014.10.120. Epub 2014 Nov 6. PMID 25500293
- See also: Click here for the Cardiothoracic Surgical Trials Network Web site. — http://www.ctsurgerynet.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mitral Valve Repair With Annuloplasty | Mitral Valve Replacement
Started | 126 | 125
Completed | 90 | 84
Not Completed | 36 | 41
Not completed — Death | 24 | 29
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Lost to Follow-up | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mitral Valve Repair With Annuloplasty | Mitral Valve Replacement | Total
Number analyzed (Participants) | 126 | 125 | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (10.2) | 67.9 (9.0) | 68.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 47 | 96
  Male | 77 | 78 | 155
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 11 | 24
  Not Hispanic or Latino | 113 | 114 | 227
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 24 | 44
  White | 104 | 98 | 202
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 25 | 26 | 51
  United States | 101 | 99 | 200

OUTCOME MEASURES:

1. Primary Outcome: Degree of Left Ventricular Remodeling, as Assessed by Left Ventricular End Systolic Volume Index (LVESVI)
Time Frame: Measured at Month 12
Measure: Mean (Standard Deviation); unit: ml per square meter of body-surface area
Arm/Group | Mitral Valve Repair With Annuloplasty | Mitral Valve Replacement
Number analyzed (Participants) | 126 | 125
ml per square meter of body-surface area | 54.6 (25.0) | 60.7 (31.5)
Statistical Analysis 1: Comparison: Mitral Valve Repair With Annuloplasty vs Mitral Valve Replacement; The trial was designed with a power of 90% to detect a between-group difference of 15 ml per square meter in the LVESVI from baseline to 12 months. We assumed a baseline LVESVI of 100 ml per square meter, improvements of 20 ml per square meter in the repair group and 35 ml per square meter in the replacement group, and equal 1-year mortality of 10 to 20% in the two groups. The primary null hypothesis was that there would be no between-group difference in the LVESVI at 12 months; Test type: Other — We tested this hypothesis in an intention-to-treat analysis using a two-tailed Wilcoxon rank-sum test, at a 0.05 alpha level. This analysis accommodated nonignorable missing LVESVI outcomes owing to the death of patients by assigning deceased patients the worst ranks in order on the basis of the time of death. We used multiple imputation for data that were missing for reasons other than death to calculate the 12-month LVESVI on the assumption that the data were missing at random; p = 0.18, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: All-cause Mortality
Time Frame: Measured at Month 24
Measure: Count of Participants; unit: Participants
Arm/Group | Mitral Valve Repair With Annuloplasty | Mitral Valve Replacement
Number analyzed (Participants) | 126 | 125
Participants | 24 | 29
Statistical Analysis 1: Comparison: Mitral Valve Repair With Annuloplasty vs Mitral Valve Replacement; Test type: Other — We used the log-rank test to compare rates of death from baseline to 2 years; p = 0.39, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.46 to 1.35]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Mitral Valve Repair With Annuloplasty | Mitral Valve Replacement
All-Cause Mortality (participants affected / at risk) | 24/126 | 29/125
Serious Adverse Events (participants affected / at risk) | 89/126 | 88/125
Other Adverse Events (participants affected / at risk) | 33/126 | 44/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitral Valve Repair With Annuloplasty (N=126) | Mitral Valve Replacement (N=125)
Bleeding (Blood and lymphatic system disorders) | 6 (7) | 10 (10)
Arrhythmias - Sustained ventricular arrhythmia (Cardiac disorders) | 10 (12) | 12 (17)
Arrhythmias - Sustained supraventricular arrhythmia (Cardiac disorders) | 23 (26) | 18 (19)
Pericardial Fluid Collection (Cardiac disorders) | 1 (1) | 1 (1)
Hepatic Dysfunction (Hepatobiliary disorders) | 5 (5) | 5 (5)
Major Infection - Localized (Infections and infestations) | 21 (25) | 21 (29)
Major Infection - Endocarditis (Infections and infestations) | 0 (0) | 2 (2)
Major Infection - Sepsis (Infections and infestations) | 11 (12) | 6 (6)
Myocardial infarction (Cardiac disorders) | 4 (5) | 1 (1)
Myocardial infarction - Peri-CABG MI (Cardiac disorders) | 0 (0) | 2 (2)
Neurological Dysfunction - TIA (Nervous system disorders) | 0 (0) | 1 (1)
Neurological Dysfunction - CVA-Ischemic (Nervous system disorders) | 8 (10) | 6 (6)
Neurological Dysfunction - CVA-Hemorrhagic (Nervous system disorders) | 2 (2) | 0 (0)
Neurological Dysfunction - Toxic Metabolic Encephalopathy (Nervous system disorders) | 2 (3) | 1 (1)
Neurological Dysfunction - Other (Nervous system disorders) | 4 (4) | 2 (2)
Renal dysfunction (no dialysis) (Renal and urinary disorders) | 4 (4) | 7 (7)
Renal failure (dialysis) (Renal and urinary disorders) | 6 (6) | 11 (11)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 18 (19)
Heart Failure (Cardiac disorders) | 30 (48) | 23 (29)
Venous Thromboembolism Event (Vascular disorders) | 4 (4) | 1 (1)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 8 (9)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Altered Mental Status (Nervous system disorders) | 1 (1) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aortic Disease (Vascular disorders) | 0 (0) | 1 (1)
Arrhythmia - Undifferentiated (Cardiac disorders) | 9 (9) | 7 (7)
Broken bone (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 6 (6)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac conduction abnormalities requiring permanent pacemaker (Cardiac disorders) | 1 (1) | 1 (1)
Carotid Disease (Vascular disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 3 (13) | 1 (1)
Coagulopathy/HIT (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Collapsed lung (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Failure to thrive (General disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
GI Bleed/GI Issue (Gastrointestinal disorders) | 9 (12) | 10 (13)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hemi-diaphragm paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxic Ischemic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Inguinal Hernia Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Left Atrial Thrombus (Cardiac disorders) | 4 (4) | 0 (0)
Orthostatic hypotension (Cardiac disorders) | 0 (0) | 1 (1)
PM or ICD Implant/Revision (Cardiac disorders) | 7 (7) | 6 (7)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Penetrating Thoracic Ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Peripheral arterial disease (Vascular disorders) | 2 (2) | 1 (1)
Re-Operation for Severe Mitral Valve Leakage (Cardiac disorders) | 0 (0) | 1 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Right Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Right groin pseudoaneurysm (Vascular disorders) | 0 (0) | 1 (1)
SIRS (General disorders) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 2 (2) | 1 (2)
Urinary retention/obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Vasoplegia (Vascular disorders) | 3 (3) | 6 (6)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Volume Overload (Cardiac disorders) | 1 (1) | 0 (0)
non-cardiac musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitral Valve Repair With Annuloplasty (N=126) | Mitral Valve Replacement (N=125)
Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmias - Sustained supraventricular arrhythmia (Cardiac disorders) | 10 (11) | 12 (12)
Hepatic Dysfunction (Hepatobiliary disorders) | 2 (2) | 3 (3)
Major Infection - Localized (Infections and infestations) | 11 (13) | 17 (21)
Myocardial infarction - Peri-Percutaneous Intervention MI (Cardiac disorders) | 1 (1) | 0 (0)
Neurological Dysfunction - Toxic Metabolic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Neurological Dysfunction - Other* (Nervous system disorders) | 0 (0) | 1 (1)
Renal dysfunction (no dialysis) (Renal and urinary disorders) | 3 (3) | 4 (4)
Renal failure (dialysis) (Renal and urinary disorders) | 2 (2) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Heart Failure (Cardiac disorders) | 2 (2) | 1 (1)
Arterial Non-CNS Thromboembolism (Vascular disorders) | 0 (0) | 1 (1)
Venous Thromboembolism Event (Vascular disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (9)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Arrhythmia - Undifferentiated (Cardiac disorders) | 0 (0) | 2 (2)
Broken bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coagulopathy/HIT (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
GI Bleed/GI Issue (Gastrointestinal disorders) | 2 (2) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Left groin lymphocele/seroma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary retention/obstruction (Renal and urinary disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes